CLINICAL TRIAL: NCT01473862
Title: Adolescent Loss: The Impact of Loss on Adolescent Oncology Patients
Acronym: ALOSS
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XPD11-150 ALOSS
Record Dates: First submitted 2011-11-08; First posted 2011-11-17 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Adolescent Oncology Patients
Keywords: adolescent; bereavement; cancer; coping skills
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Teen loss is not uncommon. Depression, emptiness, disbelief, hopelessness, and guilt are typical responses. How teens with cancer cope with the loss of a loved one or a close friend has not been well-studied in the bereavement or oncology literature. This study will describe the impact of loss on teen patients who are on treatment or have recently completed treatment for malignancy. We will look at baseline personality traits and ask teens to identify losses in their life. We will ask questions about coping and meaning-making after loss. A parent will be invited to participate -to measure parental awareness of teen loss and determine if parental coping affects teen coping. The inventories have been validated by other researchers.

DETAILED DESCRIPTION:
All participants will asked to complete a bereavement questionnaire quantifying the losses they have experienced. All participants will be screened for depression/anxiety as well as life outlook using validated tools. Patients who identify that they have experienced the loss of someone significant in their life on the bereavement questionnaire will continue with the study and complete a battery of validated psychological inventories. They will be asked to identify their most significant loss in regards to completion of the remainder of the questionnaire. In addition, those who identify losing a friend to cancer will be invited to participate in a 30-45 minute semi-structured interview (in person or via telephone) during a second session with the study staff. This interview will be audiotaped, to allow for transcription and analysis later. Parents will complete demographic information, the bereavement questionnaire, and complete inventories of family coping / cohesion regardless of child's responses to bereavement questionnaire.

In addition, those who identify losing a friend to cancer will be invited to participate in a 30-45 minute semi-structured interview (in person or via telephone) during a second session with the study staff.

Primary Objectives:

* Estimate the prevalence of loss, with particular interest in the extent of peer loss, in adolescent oncology patients who have been on therapy ≥ 12 months (≥ 6 months if progressive or refractory disease) or off therapy for ≤ 3 years.
* Describe the impact of loss on adolescent oncology patients by focusing on coping efficacy, psychological distress, meaning-making, and complicated bereavement.

Secondary Objective:

* Describe parental knowledge of losses experienced by an adolescent child who has recently undergone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-21 inclusive at time of study enrollment
* English speaking
* Research participant carries a diagnosis of a malignancy (or serious non-malignant disorder requiring HSCT) >12 months.
* Research participant carries a diagnosis of a malignancy (or serious non-malignant disorder requiring HSCT) for >6 months and <12 months but has evidence of refractory/progressive disease.
* Patients who have completed cancer-directed therapy >36 months ago are not eligible. (Note: Allogenic transplant recipients will be considered "off-therapy" 1 year after HSCT.)
* No known history of significant cognitive deficits (i.e. with major impairments) that would preclude completion of study measures; not meant to exclude research participants with mild learning problems.
* Research participant and 1 parent willing to participate and provide consent/assent according to institutional guidelines. Parent may decline to participate in parental inventories, but consent to adolescent participation.

Exclusion Criteria:

* Less than 13-years of age at completion of therapy.
* Patients on hospice who are without scheduled follow-up at St. Jude Children's Research Hospital (SJCRH)
* "Observation" patients. Patients that are being followed by imaging due to previous identification of an atypical lesion on radiographic imaging not identified to have a specific diagnosis.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: English-speaking adolescent oncology patients (age 13-21) at St. Jude Children's Research Hospital who have been on therapy for ≥ 12 months (≥ 6 months if progressive or refractory disease) OR off therapy for ≤ 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants who have experienced the death of a friend or relative by type of loss. | Once on Day 1
  The prevalence of loss among the participants will be calculated. The type of losses will be described.
Descriptive statistics of coping efficacy scores, psychological distress scores, meaning-making scores, and complicated bereavement scores. | Once on Day 1
  All data for this objective will be mainly analyzed in a descriptive manner. The score for coping efficacy will be calculated from the General Coping Efficacy instrument. In addition, a subset of participants who identify losing a friend to cancer will be invited to complete a 30-45 minute semi-structured interview.

SECONDARY OUTCOMES:
Number of parents with knowledge of losses experienced by adolescent child. | Once on Day 1
  Descriptive analysis from the Bereavement Questionnaire (parent version).

CONTACTS AND LOCATIONS:
Overall Officials: Liza Johnson, MD,MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols